CLINICAL TRIAL: NCT01089127
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Different Doses of Indacaterol in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease, Using Salmeterol as an Active Control
Brief Title: Efficacy and Safety of Different Doses of Indacaterol in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2356
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Indacaterol; COPD; salmeterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Indacaterol 18.75 μg (Experimental): Patients inhaled indacaterol 18.75 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to salmeterol
- Indacaterol 37.5 μg (Experimental): Patients inhaled indacaterol 37.5 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to salmeterol
- Indacaterol 75 μg (Experimental): Patients inhaled indacaterol 75 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to salmeterol
- Indacaterol 150 μg (Experimental): Patients inhaled indacaterol 150 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to salmeterol
- Salmeterol 50 μg (Active Comparator): Patients inhaled salmeterol 50 μg twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. In addition, patients inhaled placebo to indacaterol once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
  Interventions: Drug: Salmeterol 50 μg; Drug: Placebo to indacaterol
- Placebo (Placebo Comparator): Patients inhaled placebo to indacaterol once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
  Interventions: Drug: Placebo to indacaterol; Drug: Placebo to salmeterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Indacaterol 150 μg; Indacaterol 18.75 μg; Indacaterol 37.5 μg; Indacaterol 75 μg
Drug: Salmeterol 50 μg — Salmeterol was supplied in the manufacturer's proprietary Diskus inhaler device.
  Arms: Salmeterol 50 μg
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Placebo; Salmeterol 50 μg
Drug: Placebo to salmeterol — Placebo to salmeterol was supplied in the manufacturer's proprietary Diskus inhaler device.
  Arms: Indacaterol 150 μg; Indacaterol 18.75 μg; Indacaterol 37.5 μg; Indacaterol 75 μg; Placebo

SUMMARY:
This study compared the 14-day bronchodilator efficacy of indacaterol with that of placebo and salmeterol.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease [GOLD] Guidelines, 2008) and:

  1. Smoking history of at least 10 pack-years
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value
  3. Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion criteria:

* Patients who have had a COPD exacerbation requiring systemic corticosteroids and/or antibiotics and/or hospitalization in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (67):
  - Novartis Investigator Site, Florence, Alabama
  - Novartis Investigator Site, Jasper, Alabama
  - Novartis Investigator Site, Phoenix, Arizona
  - Novartis Investigator Site, Searcy, Arkansas
  - Novartis Investigator Site, Fullerton, California
  - Novartis Investigative Site, Rancho Mirage, California
  - Novartis Investigator Site, Riverside, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, Stockton, California
  - Novartis Investigator Site, Temecula, California
  - Novartis Investigator Site, Walnut Creek, California
  - Novartis Investigator Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Glastonbury, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigator Site, Clearwater, Florida
  - Novartis Investigator Site, DeFuniak Springs, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigator Site, Miami, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigator Site, Tampa, Florida
  - Novartis Investigator Site, O'Fallon, Illinois
  - Novartis Investigator Site, Florence, Kentucky
  - Novartis Investigator Site, Madisonville, Kentucky
  - Novartis Investigator Site, Opelousas, Louisiana
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigator Site, Edina, Minnesota
  - Novartis Investigator Site, Fridley, Minnesota
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Ozark, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Bellevue, Nebraska
  - Novartis Investigator Site, Lincoln, Nebraska
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Henderson, Nevada
  - Novartis Investigator Site, Las Vegas, Nevada
  - Novartis Investigator Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Cherry Hill, New Jersey
  - Novartis Investigative Site, Bayside, New York
  - Novartis Investigative Site, Great Neck, New York
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, Larchmont, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigator Site, Cadiz, Ohio
  - Novartis Investigator Site, Canton, Ohio
  - Novartis Investigator Site, Columbus, Ohio
  - Novartis Investigator Site, Toledo, Ohio
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigator Site, Medford, Oregon
  - Novartis Investigative Site, Phoenixville, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative site, Charleston, South Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Easley, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigator Site, Cookeville, Tennessee
  - Novartis Investigator Site, Dickinson, Texas
  - Novartis Investigator Site, Fort Worth, Texas
  - Novartis Investigator Site, McKinney, Texas
  - Novartis Investigator Site, Salt Lake City, Utah
  - Novartis Investigative Site, Fredericksburg, Virginia
  - Novartis Investigative site, Newport News, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigator Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 18.75 μg | Indacaterol 37.5 μg | Indacaterol 75 μg | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Started | 92 | 91 | 94 | 92 | 92 | 91
Exposed to Study Drug | 89 (3 randomized patients in this group were not exposed to study treatment.) | 90 (1 randomized patient in this group was not exposed to study treatment.) | 94 | 92 | 91 (1 randomized patient in this group was not exposed to study treatment.) | 91
Completed | 84 | 86 | 92 | 91 | 90 | 88
Not Completed | 8 | 5 | 2 | 1 | 2 | 3
Not completed — Adverse Event | 5 | 1 | 1 | 0 | 0 | 1
Not completed — Subject withdrew consent | 0 | 1 | 1 | 1 | 0 | 2
Not completed — Abnormal test procedure result(s) | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 18.75 μg | Indacaterol 37.5 μg | Indacaterol 75 μg | Indacaterol 150 μg | Salmeterol 50 μg | Placebo | Total
Number analyzed (Participants) | 89 | 90 | 94 | 92 | 91 | 91 | 547
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures are based on safety population. 3 patients in the indacaterol 18.75 ug group, 1 patient in the indacaterol 37.5 ug group, and 1 patient in the salmeterol 50 ug group were randomized but were not exposed to study treatment and were not included in the calculation of demographic data.
  years | 62.8 (8.95) | 61.9 (9.61) | 62.6 (9.30) | 62.3 (9.50) | 62.4 (9.52) | 63.6 (8.44) | 62.6 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 40 | 39 | 47 | 43 | 251
  Male | 50 | 47 | 54 | 53 | 44 | 48 | 296

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of the Study (Week 2 + 1 Day, Day 15)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose at the end of the study (Week 2 + 1 day, Day 15)
Population: Full analysis set: All randomized patients who received at least 1 dose of study drug, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 18.75 μg | Indacaterol 37.5 μg | Indacaterol 75 μg | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Number analyzed (Participants) | 82 | 84 | 87 | 90 | 88 | 86
Liters | 1.35 (0.020) | 1.38 (0.019) | 1.38 (0.019) | 1.40 (0.019) | 1.39 (0.019) | 1.28 (0.019)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose on Day 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose on Day 2. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose on Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 18.75 μg | Indacaterol 37.5 μg | Indacaterol 75 μg | Indacaterol 150 μg | Salmeterol 50 μg | Placebo
Number analyzed (Participants) | 85 | 86 | 88 | 91 | 88 | 86
Liters | 1.33 (0.015) | 1.34 (0.015) | 1.38 (0.015) | 1.40 (0.014) | 1.41 (0.015) | 1.28 (0.015)

ADVERSE EVENTS:
Description: Safety population.
Groups:
- Indacaterol 18.75 ug: Patients inhaled indacaterol 18.75 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
- Indacaterol 37.5 ug: Patients inhaled indacaterol 37.5 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
- Indacaterol 75 ug: Patients inhaled indacaterol 75 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
- Indacaterol 150 ug: Patients inhaled indacaterol 150 μg once daily in the morning via the Concept1 single-dose dry-powder inhaler (SDDPI). In addition, patients inhaled placebo to salmeterol twice daily, once in the morning and once in the evening, via the manufacturer's proprietary Diskus inhaler. Treatment continued for 2 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. Albuterol via a multi-dose dry-powder inhaler (MDI) was available for rescue use throughout the study.
Arm/Group | Indacaterol 18.75 ug | Indacaterol 37.5 ug | Indacaterol 75 ug | Indacaterol 150 ug | Salmeterol 50 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/89 | 0/90 | 0/94 | 1/92 | 0/91 | 3/91
Other Adverse Events (participants affected / at risk) | 1/89 | 7/90 | 8/94 | 2/92 | 4/91 | 9/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 18.75 ug (N=89) | Indacaterol 37.5 ug (N=90) | Indacaterol 75 ug (N=94) | Indacaterol 150 ug (N=92) | Salmeterol 50 μg (N=91) | Placebo (N=91)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 18.75 ug (N=89) | Indacaterol 37.5 ug (N=90) | Indacaterol 75 ug (N=94) | Indacaterol 150 ug (N=92) | Salmeterol 50 μg (N=91) | Placebo (N=91)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 7 | 1 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.